CLINICAL TRIAL: NCT01229852
Title: Treatment of Fibromyalgia Using Deep Shaped-Field (DSF) Transcranial Magnetic Stimulation (TMS): A Clinical Feasibility Study
Brief Title: Treatment of Fibromyalgia Using Deep Shaped-Field Transcranial Magnetic Stimulation a Clinical Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cervel Neurotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-CFS-FM-1
Record Dates: First submitted 2010-10-25; First posted 2010-10-28 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Transcranial Magnetic Stimulation; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active DSF-rTMS (Experimental): Active rTMS treatment.
  Interventions: Device: DSF-rTMS

INTERVENTIONS:
Device: DSF-rTMS — Effective Transcranial Magnetic Stimulation

SUMMARY:
Deep shaped-field transcranial magnetic stimulation is a new type of transcranial magnetic stimulation technology which may provide a drug-free method for treating fibromyalgia.

The purpose of this study is to determine the effectiveness and the durability of effect of Deep shaped-field repetitive transcranial magnetic stimulation (rTMS) in men and women diagnosed with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia as diagnosed by American College of Rheumatology (ACR) criteria.
* Moderate or severe pain from fibromyalgia despite current treatment regimen.
* Will not become pregnant during study.

Exclusion Criteria:

* Seizure disorder.
* Metal implants on or in brain, spinal cord, ear, eye or heart.
* Current use of proconvulsant medications (e.g., bupropion).
* Taking oral amitriptyline > 100 mg once daily at bedtime.
* Nonscheduled analgesic, anticonvulsant or antidepressant medications.
* Severe depression or suicidality.
* Other significant psychiatric disorder.
* Previous use of TMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on the Brief Pain Inventory (BPI) | Daily during 20 day treatment

SECONDARY OUTCOMES:
Change from Baseline on the Beck Depression Inventory Second Edition (BDI-II) | 1, 6, 10, 15 day of treatment; 1 day, 4 weeks post treatment
Change from Baseline for the Fibromyalgia Impact Questionnaire (FIQ) | 1, 10 day of treatment; 1 day and 4 weeks post treatment
Durability, safety and tolerability | Measured weekly up to 1 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: M. Bret Schneider, M.D., Study Chair — Cervel Neurotech, Inc.
Locations (1):
- Premier Research Group, Phoenix, Arizona, United States

REFERENCES:
- See also: Cervel Neurotech, Inc. Homepage — http://www.cervel.com